CLINICAL TRIAL: NCT03531385
Title: Assessment of Central Sensitization, Neuropathic Pain, Sleep Quality and Daily Life Activities in Behcet's Disease and Healthy Controls
Brief Title: Assessment of Central Sensitization, Neuropathic Pain, Sleep Quality and Daily Life Activities in Behcet's Disease
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Koray Ayar, Assistant Professor, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-25 2018/03-12
Record Dates: First submitted 2018-05-09; First posted 2018-05-21 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Behcet's Disease; Central Sensitisation
Keywords: Behcet's disease; Central sensitisation; Neuropathic pain; Sleep disturbance
MeSH Terms: conditions — Behcet Syndrome; Neuralgia; Parasomnias | interventions — Central Nervous System Sensitization; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Behcet: Patients diagnosed with Behcet disease
  Interventions: Diagnostic Test: Central sensitisation; Diagnostic Test: Neuropathic pain; Other: Sleep disturbance; Other: Quality of life
- Healthy controls: Individuals without any chronic disease
  Interventions: Diagnostic Test: Central sensitisation; Diagnostic Test: Neuropathic pain; Other: Sleep disturbance; Other: Quality of life

INTERVENTIONS:
Diagnostic Test: Central sensitisation — Central Sensitization Inventory, which is a comprehensive self-report inventory to assess the overlapping symptom dimensions of central sensitisation syndrome will be used to identify participants with central sensitisation.
Diagnostic Test: Neuropathic pain — Frequency of neuropatic pain will be investigated using Pain Detect Questionnaire
Other: Sleep disturbance — Assessment of sleep disturbance will be assessed by Pittsburgh Sleep Quality Index
Other: Quality of life — Quality of life will be assessed by the Nottingham Health Profile

SUMMARY:
There are few studies in the literature regarding increased frequency of neuropathic pain and sleep disturbance and decreased quality of life in Behçet's disease. Frequency of central sensitization was not investigated in patients with Behçet's disease before. In this study, it is aimed to investigate the frequency of central sensitization, neuropathic pain, sleep disorder and quality of life and their relation to each other in Behcet's disease.

DETAILED DESCRIPTION:
Central sensitization reduces the pain threshold in the pain pathways of the nervous system, causing pain sensation to be perceived with lower stimuli and often causing chronic pain. Central sensitization can be seen with many conditions such as neuropathic pain and sleep disorders, as well as with inflammatory diseases such as rheumatoid arthritis. There are few studies in the literature regarding increased frequency of neuropathic pain and sleep disturbance and decreased quality of life in Behçet's disease. Frequency of central sensitization was not investigated in patients with Behçet's disease before. In this study, it is aimed to investigate the frequency of central sensitization, neuropathic pain, sleep disorder and quality of life and their relation to each other in patients with Behcet's disease and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Behcet disease according to international study group criteria
* Healthy volunteers without previously known systemic chronic disease
* Patients older than 18
* Patients younger than 75

Exclusion Criteria:

* Participants which were previously diagnosed with diabetes mellitus
* Participants which were previously diagnosed with chronic renal failure
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population consists of participants who are between age 18-75, not pregnant and who were not diagnosed previously with diabetes mellitus or chronic renal failure
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Central Sensitisation Inventory | 6 months
  A self-report inventory, the Central Sensitization Inventory (CSI), will be used to assess the overlapping symptom dimensions of Central Sensitivity Syndromes. This measure is intended as a screening instrument to help identify the presence of a Central Sensitivity Syndrome, and to alert clinicians that presenting symptoms may be related to central sensitisation. Part A of the Central Sensitisation Inventory assesses 25 health-related symptoms that are common to Central Sensitivity Syndrome, with total scores ranging from 0-100. Part B (which is not scored) asks if one has previously been diagnosed with one or more specific disorders, including seven separate Central Sensitivity Syndromes

SECONDARY OUTCOMES:
Pain Detect Questionaire | 6 months
  The pain detect questionnaire was specifically developed to detect neuropathic pain components in adult patients. The questionnaire consists of seven questions that address the quality of neuropathic pain symptoms; it is completed by the patient and no physical examination is required. The first five questions ask about the gradation of pain, scored from 0 to 5 (never = 0, hardly noticed = 1, slightly = 2; moderately = 3, strongly = 4, very strongly = 5). Question 6 asks about the pain course pattern, scored from -1 to 2, depending on which pain course pattern diagram is selected. Question 7 asks about radiating pain, answered as yes or no, and scored as 2 or 0 respectively. The final score between -1 and 38, indicates the likelihood of a neuropathic pain component. A score of <13 indicates that pain is unlikely to have a neuropathic component (< 15%), while a score of 19 < suggests that pain is likely to have a neuropathic component (> 90%).
Pittsburgh Sleep Quality Index | 6 months
  It is composed of 19 questions, which create 7 major components. Each component is scored from 0 to 3 points, in which lower point denotes no problems, while higher score denotes worsening problems in following order: (1) subjective sleep quality (very good vs. very bad), (2) sleep latency (≤15 min to >60 min), (3) sleep duration (≥7 h to <5 h), (4) sleep efficiency (≥85% to <65% h sleep/hours in bed), (5) sleep disturbances (not during the past month to ≥3 times per week), (6) use of sleeping medications (none to ≥3 times a week) and (7) daytime dysfunction (not a problem to a very big problem). All 7 components are then summed up to create a scale from 0 to 21 points.
Nottingham Health Profile | 6 months
  Health related quality of life of the patients was evaluated with the Nottingham Health Profile, which contains 38 items in 6 domains related to level of energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), physical mobility (8 items), and social isolation (5 items). Items in each domain are assigned a weight; the total score for each domain is 100; a score of 0 indicates good subjective health status, while 100 indicates poor subjective health status. Total Nottingham Health Profile total score is obtained by averaging the 6 domain scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Education and Research Hospital, Bursa, Turkey (Türkiye)